CLINICAL TRIAL: NCT01689519
Title: A Phase III, Double-Blind, Placebo-Controlled Study of Vemurafenib Versus Vemurafenib Plus GDC-0973 in Previously Untreated BRAF^600-Mutation Positive Patients With Unresectable Locally Advanced or Metastatic Melanoma
Brief Title: A Study Comparing Vemurafenib Versus Vemurafenib Plus Cobimetinib in Participants With Metastatic Melanoma
Acronym: coBRIM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GO28141; 2012-003008-11 (EudraCT Number)
Record Dates: First submitted 2012-09-18; First posted 2012-09-21 (Estimated); Results first posted 2015-10-30 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Malignant Melanoma
Keywords: Zelboraf; vemurafenib; RG7204; PLX4032; Genentech MEK inhibitor; Genentech BRAF inhibitor; Roche MEK inhibitor; Roche BRAF inhibitor; RO5185426; metastatic melanoma; BRAF positive melanoma; BRAF mutant melanoma; advanced melanoma; Genentech RAF inhibitor; Roche RAF inhibitor; BRAF V600E kinase inhibitor; Oncogenic BRAF inhibitor; BRAF kinase inhibitor; GDC-0973; XL518; melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Placebo + Vemurafenib (Active Comparator): Participants will receive placebo orally once daily on Days 1-21 of each 28-day cycle plus vemurafenib 960 milligrams (mg) orally twice a day on Days 1-28 of each 28-day cycle until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurs earliest.
  Interventions: Drug: Placebo; Drug: Vemurafenib
- Cobimetinib + Vemurafenib (Experimental): Participants will receive cobimetinib 60 mg orally once daily on Days 1-21 of each 28-day cycle plus vemurafenib 960 mg orally twice a day on Days 1-28 of each 28-day cycle until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurs earliest.
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib

INTERVENTIONS:
Drug: Placebo — Placebo supplied as tablets
  Arms: Placebo + Vemurafenib
Drug: Vemurafenib — Vemurafenib supplied as tablets
  Other Names: RO518426
Drug: Cobimetinib — Cobimetinib supplied as tablets
  Other Names: GDC-0973; RO5514041; XL518
  Arms: Cobimetinib + Vemurafenib

SUMMARY:
To evaluate the efficacy of vemurafenib in combination with cobimetinib (GDC-0973), compared with vemurafenib and placebo, in previously untreated BRAF V600 mutation-positive patients with unresectable locally advanced or metastatic melanoma, as measured by progression-free survival (PFS), assessed by the study site investigator.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed melanoma, either unresectable stage IIIc or stage IV metastatic melanoma, as defined by the American Joint Committee on Cancer 7th edition. Unresectability of stage IIIc disease must have confirmation from a surgical oncologist
* Participants must be naïve to treatment for locally advanced unresectable or metastatic disease (ie, no prior systemic anti-cancer therapy for advanced disease; stage IIIc and IV). Prior adjuvant immunotherapy (including ipilimumab) is allowed
* Documentation of BRAF V600 mutation-positive status in melanoma tumor tissue (archival or newly obtained tumor samples) using the cobas 4800 BRAF V600 mutation test
* Measurable disease per RECIST v1.1
* Eastern Clinical Oncology Group performance status of 0 or 1
* Consent to provide archival for biomarker analyses
* Consent to undergo tumor biopsies for biomarker analyses
* Life expectancy greater than or equal to (≥) 12 weeks
* Adequate hematologic and end organ function

Exclusion Criteria:

* History of prior rapidly accelerated fibrosarcoma or mitogen-activated protein kinase pathway inhibitor treatment
* Palliative radiotherapy within 14 days prior to the first dose of study treatment
* Major surgery or traumatic injury within 14 days prior to first dose of study treatment
* Active malignancy other than melanoma that could potentially interfere with the interpretation of efficacy measures. Participants with a previous malignancy within the past 3 years are excluded except for participants with resected basal cell carcinoma or squamous cell carcinoma of the skin, melanoma in-situ, carcinoma in-situ of the cervix, and carcinoma in-situ of the breast
* History of or evidence of retinal pathology on ophthalmological examination that is considered a risk factor for neurosensory retinal detachment, retinal vein occlusion, or neovascular macular degeneration
* Uncontrolled glaucoma with intraocular pressure
* Serum cholesterol ≥ Grade 2
* Hypertriglyceridemia ≥ Grade 2
* Hyperglycemia (fasting) ≥ Grade 2
* History of clinically significant cardiac dysfunction
* Participants with active central nervous system (CNS) lesions (including carcinomatous meningitis) are excluded. However, participants are eligible if:

  1. All known CNS lesions have been treated with stereotactic therapy or surgery, AND
  2. There has been no evidence of clinical and radiographic disease progression in the CNS for ≥ 3 weeks after radiotherapy or surgery
* Current severe, uncontrolled systemic disease
* History of malabsorption or other condition that would interfere with absorption of study drugs
* Pregnant, lactating, or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2014-05-09 (Actual); Study Completion 2019-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (156):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - The Angeles Clinic and Research Institute - W LA Office, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - University Of Colorado, Aurora, Colorado
  - Florida Cancer Specialists - Broadway, Fort Myers, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Inc., Orlando, Florida
  - Northwestern Center For Clinical Research, Chicago, Illinois
  - Uni of Kansas Medical Center; Dept of Neurology, Kansas City, Kansas
  - U of L - Physicians Pulmonology; Dept of Neuroradiology and Dept of Diagnostic Radiology, Louisville, Kentucky
  - Washington University School of Medicine; Dept of Medicine/Div of Medical Oncology, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center; Department of Medicine, Lebanon, New Hampshire
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - St. Luke's University Health network, Bethlehem, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital; Investigational Services, Providence, Rhode Island
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (17):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Lismore Base Hospital; Cancer Care & Haematology Unit, Lismore, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, New South Wales
  - Royal Darwin Hospital, Casuarina, Northern Territory
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Royal Adelaide Hospital; Hepatology, Adelaide, South Australia
  - Ashford Cancer Centre, Ashford SA, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Launceston General Hospital; Gastroenterology Research, Launceston, Tasmania
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre-East Melbourne, Melbourne, Victoria
  - The Alfred Hospital, Prahan, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (3):
  - Ordensklinikum Linz Elisabethinen, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
  - Medizinische Universität Wien, Vienna
- Belgium (6):
  - Institut Jules Bordet; Department of Medical Oncology, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Antwerpen, Edegem
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - CHU Sart-Tilman, Liège
  - AZ Delta (Campus Rumbeke), Roeselare
- Canada (7):
  - BC Cancer Agency Vancouver Island Cancer Centre, Victoria, British Columbia
  - Juravinski Cancer Clinic; Department of Oncology, Hamilton, Ontario
  - The Ottawa Hospital Cancer Center; General Campus, Ottawa, Ontario
  - Toronto Sunnybrook Hospital, Toronto, Ontario
  - Princess Margaret Hospital; Department of Med Oncology, Toronto, Ontario
  - London Health Sciences Centre · Victoria Hospital;Department of Pediatrics, London, Quebec
  - McGill University Health Centre/Glen Site / Royal Victoria Hospital, Montreal, Quebec
- Czechia (9):
  - Masarykuv onkologicky ustav, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Multiscan s.r.o., Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Fakultni nemocnice Motol; Neurologicka klinika, Prague
  - Nemocnice Na Bulovce, Prague
- France (13):
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux
  - Hôpital Ambroise Paré - Boulogne-Billancourt; Respiratory, Boulogne-Billancourt
  - CHU Clermont Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - CHU de Dijon - Hopital le Bocage, Dijon
  - Centre Hospitalier Universitaire de Grenoble - Albert Michallon, La Tronche
  - Hopital Claude Huriez - CHU Lille, Lille
  - Hopital de la Timone, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU NANTES - Hôtel Dieu; Pharmacy, Nantes
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Robert Debre; DERMATOLOGIE, Reims
  - Centre Eugene Marquis; Service d'oncologie, Rennes
- Germany (20):
  - St. Josef-Hospital; Studienambulanz, Bochum
  - Elbekliniken Buxtehude GmbH, Buxtehude
  - Universitaetsklinikum Koeln; Hematology/Oncology, Cologne
  - Universitätsklinikum "Carl Gustav Carus" der Technischen Universität Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Essen, Essen
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - SRH Wald-Klinikum Gera; Klinik für Hautkrankheiten und Allergologie, Gera
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel; Klinik fuer Allgemeine Innere Medizin, Kiel
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Klinikum der Ludwigs-Maximilians-Universitaet Muenchen, München
  - Fachklinik Hornheide, Münster
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Wurzburg, Würzburg
- Hungary (4):
  - Orszagos Onkologiai Intezet, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Pécs
  - Szegedi Tud.Egyetem Szent-Gyorgyi Albert Klin.Kozp., Szeged
- Israel (6):
  - Soroka Medical Center; Oncology Dept, Beersheba
  - Rambam Health Care Campus, Haifa
  - HADASSAH UNIVERSITY HOSPITAL, EIN KAREM; Oncology, Jerusalem
  - Rabin Medical Center-Beilinson Campus;Hematology-Oncology, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky MC, Dana children's hospital;Oncology Division, Tel Aviv
- Italy (11):
  - Istituto Tumori Giovanni Paolo II IRCSS; Ospedale Oncologico Bari, Bari, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori, Meldola, Emilia-Romagna
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Istituto Nazionale Tumori Regina Elena IRCCS, Rome, Lazio
  - Istituto Nazionale per la Ricerca sul Cancro di Genova, Genoa, Liguria
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII (Presidio Papa Giovanni XXIII), Bergamo, Lombardy
  - Asst Degli Spedali Civili Di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - A.O.U. Senese Policlinico Santa Maria Alle Scotte, Siena, Tuscany
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Veneto
- Netherlands (3):
  - Amsterdam UMC Location VUMC, Amsterdam
  - Leids Universitair Medisch Centrum; Cardiology, Leiden
  - Maastricht University Medical Center, Maastricht
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Waikato Hospital, Hamilton
- Radiumhospitalet, Oslo, Norway
- Russia (5):
  - TSBHI Altai Territorial oncological dispensary, Barnaul
  - FSBSI "N. N. Blokhin Russian Cancer Research Center", Moscow
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - Pyatigorsky Oncologic Dispensary, Pyatigorsk
- Spain (8):
  - Complexo Hospitalario Universitario de Santiago, Santiago de Compostela, LA Coruña
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (4):
  - Länssjukhuset Ryhov, Jönköping
  - Skånes Universitetssjukhus, Lund
  - Sahlgrenska Sjukhuset, Mölnlycke
  - Akademiska Sjukhuset, Uppsala
- Switzerland (2):
  - Inselspital-Universitaetsspital Bern, Bern
  - Kantonsspital Graubuenden, Chur
- United Kingdom (15):
  - Bristol Haematology and Oncology Centre, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Beatson West of Scotland Cancer Centre, Glasgow
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts and the London NHS Trust., London
  - St George's Hospital; Courtyard Clinic, London
  - Royal Marsden Hospital - Fulham, London
  - Royal Marsden Hospital - London, London
  - Freeman Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals; QMC Campus, Nottingham
  - Southampton General Hospital, Southampton
  - Royal Cornwall Hospital, Truro
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Barteselli G, Goodman GR, Patel Y, Caro I, Xue C, McCallum S. Characterization of Serous Retinopathy Associated with Cobimetinib: Integrated Safety Analysis of Four Studies. Drug Saf. 2022 Dec;45(12):1491-1499. doi: 10.1007/s40264-022-01248-2. Epub 2022 Oct 30. PMID 36310331
- [Derived] Ascierto PA, Dreno B, Larkin J, Ribas A, Liszkay G, Maio M, Mandala M, Demidov L, Stroyakovskiy D, Thomas L, de la Cruz-Merino L, Atkinson V, Dutriaux C, Garbe C, Hsu J, Jones S, Li H, McKenna E, Voulgari A, McArthur GA. 5-Year Outcomes with Cobimetinib plus Vemurafenib in BRAFV600 Mutation-Positive Advanced Melanoma: Extended Follow-up of the coBRIM Study. Clin Cancer Res. 2021 Oct 1;27(19):5225-5235. doi: 10.1158/1078-0432.CCR-21-0809. PMID 34158360
- [Derived] Ascierto PA, Ribas A, Larkin J, McArthur GA, Lewis KD, Hauschild A, Flaherty KT, McKenna E, Zhu Q, Mun Y, Dreno B. Impact of initial treatment and prognostic factors on postprogression survival in BRAF-mutated metastatic melanoma treated with dacarbazine or vemurafenib +/- cobimetinib: a pooled analysis of four clinical trials. J Transl Med. 2020 Aug 3;18(1):294. doi: 10.1186/s12967-020-02458-x. PMID 32746839
- [Derived] de la Cruz-Merino L, Di Guardo L, Grob JJ, Venosa A, Larkin J, McArthur GA, Ribas A, Ascierto PA, Evans JTR, Gomez-Escobar A, Barteselli G, Eng S, Hsu JJ, Uyei A, Dreno B. Clinical features of serous retinopathy observed with cobimetinib in patients with BRAF-mutated melanoma treated in the randomized coBRIM study. J Transl Med. 2017 Jun 24;15(1):146. doi: 10.1186/s12967-017-1246-0. PMID 28646893
- [Derived] Dreno B, Ribas A, Larkin J, Ascierto PA, Hauschild A, Thomas L, Grob JJ, Koralek DO, Rooney I, Hsu JJ, McKenna EF, McArthur GA. Incidence, course, and management of toxicities associated with cobimetinib in combination with vemurafenib in the coBRIM study. Ann Oncol. 2017 May 1;28(5):1137-1144. doi: 10.1093/annonc/mdx040. PMID 28444112
- [Derived] Ascierto PA, McArthur GA, Dreno B, Atkinson V, Liszkay G, Di Giacomo AM, Mandala M, Demidov L, Stroyakovskiy D, Thomas L, de la Cruz-Merino L, Dutriaux C, Garbe C, Yan Y, Wongchenko M, Chang I, Hsu JJ, Koralek DO, Rooney I, Ribas A, Larkin J. Cobimetinib combined with vemurafenib in advanced BRAF(V600)-mutant melanoma (coBRIM): updated efficacy results from a randomised, double-blind, phase 3 trial. Lancet Oncol. 2016 Sep;17(9):1248-60. doi: 10.1016/S1470-2045(16)30122-X. Epub 2016 Jul 30. PMID 27480103
- [Derived] Larkin J, Ascierto PA, Dreno B, Atkinson V, Liszkay G, Maio M, Mandala M, Demidov L, Stroyakovskiy D, Thomas L, de la Cruz-Merino L, Dutriaux C, Garbe C, Sovak MA, Chang I, Choong N, Hack SP, McArthur GA, Ribas A. Combined vemurafenib and cobimetinib in BRAF-mutated melanoma. N Engl J Med. 2014 Nov 13;371(20):1867-76. doi: 10.1056/NEJMoa1408868. Epub 2014 Sep 29. PMID 25265494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Written informed consent for participation in the study was obtained before performing any study-specific screening tests or evaluations.
Groups:
- Cobimetinib + Vemurafenib: Participants received cobimetinib 60 mg orally once daily on Days 1-21 of each 28 day cycle plus vemurafenib 960 mg orally twice a day on Days 1-28 of each 28 day cycle until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurs earliest.
- Placebo + Vemurafenib: Participants received placebo orally once daily on Days 1-21 of each 28 day cycle plus vemurafenib 960 mg orally twice a day on Days 1-28 of each 28 day cycle until disease progression, death, unacceptable toxicity, or withdrawal of consent, whichever occurs earliest.
Period: Intent to Treat
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Started | 247 | 248
Completed | 0 | 0
Not Completed | 247 | 248
Not completed — Death | 157 | 167
Not completed — Lost to Follow-up | 4 | 8
Not completed — Other | 2 | 4
Not completed — Physician Decision | 4 | 1
Not completed — Study terminated by Spon6sor | 59 | 48
Not completed — Withdrawal by Subject | 21 | 20
Period: Safety Population
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Started | 248 | 245
Completed | 0 | 0
Not Completed | 248 | 245
Not completed — Death | 158 | 165
Not completed — Lost to Follow-up | 4 | 8
Not completed — Other | 2 | 4
Not completed — Physician Decision | 4 | 1
Not completed — Study Terminated By Sponsor | 60 | 47
Not completed — Withdrawal by Subject | 20 | 20

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants, regardless of whether or not study treatment was received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib | Total
Number analyzed (Participants) | 247 | 248 | 495
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 179 | 362
  >=65 years | 64 | 69 | 133
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.9 (14.0) | 55.3 (13.8) | 55.1 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 108 | 209
  Male | 146 | 140 | 286
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Asian | 1 | 0 | 1
  More than one race | 1 | 1 | 2
  Native Hawaiian or other Pacific Islande | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 227 | 235 | 462
  Unknown or Not Reported | 16 | 9 | 25
  Other | 2 | 2 | 4
Race/Ethnicity, Customized [Number; unit: Count of Participants]
  Hispanic or Latino | 14 | 12 | 26
  Not Hispanic or Latino | 213 | 223 | 436
  Not Stated | 16 | 10 | 26
  Unknown | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from randomization to the first occurrence of disease progression, as determined by the investigator using Response Evaluation Criteria in Solid Tumors v1.1, or death from any cause, whichever came first. Disease progression was defined as: (1) at least a 20% increase in the sum (the increase in the sum must be at least 5 mm) of diameters of target lesions, taking as reference the smallest sum during the study; (2) unequivocal progression of existing non-target lesions; or (3) the appearance of 1 or more new lesions.
Time Frame: Baseline to the 21 July 2019 data cut-off (up to 7 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Number analyzed (Participants) | 247 | 248
Months
  Primary Analysis: 9 May 2014 | 9.90 [9.00 to NA] — NA = not estimable, could not be calculated due to too few events. | 6.20 [5.55 to 7.39]
  Post hoc Efficacy Analysis: 16 January 2015 | 12.30 [9.50 to 13.40] | 7.20 [5.60 to 7.50]
  Extended 5-Year Analysis: 21 July 2019 | 12.60 [9.50 to 14.80] | 7.20 [5.60 to 7.50]
Statistical Analysis 1: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Primary Analysis 9 May 2014; Test type: Superiority or Other; p = 0.0001, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.39 to 0.68]
Statistical Analysis 2: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Post hoc Efficacy Analysis: 16 January 2015; Test type: Superiority or Other; p < 0.0001, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.46 to 0.72]
Statistical Analysis 3: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Extended 5-Year Analysis: 21 July 2019; Test type: Superiority or Other; p < 0.0001, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.53 to 0.79]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from randomization until the date of death from any cause.
Time Frame: Baseline to the 21 July 2019 data cut-off (up to 7 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether or not study treatment was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Number analyzed (Participants) | 247 | 248
Months
  Primary Analysis 9 May 2014 | NA [NA to NA] — NA = not estimable, could not be calculated due to too few events. | NA [NA to NA] — NA = not estimable, could not be calculated due to too few events.
  Post hoc Analysis 16 January 2015 | NA [20.70 to NA] — NA = not estimable, could not be calculated due to too few events. | 17.00 [15.00 to NA] — NA = not estimable, could not be calculated due to too few events.
  Final Analysis 28 August 2015 | 22.30 [20.3 to NA] — NA = not estimable, could not be calculated due to too few events. | 17.40 [15.00 to 19.8]
  Extended 5-year Analysis 21 July 2019 | 22.50 [20.30 to 28.80] | 17.40 [15.00 to 19.80]
Statistical Analysis 1: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Primary Analysis 9 May 2014; Test type: Superiority or Other; p = 0.0463, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.645, 95% CI 2-sided [0.42 to 1.00]
Statistical Analysis 2: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Post hoc Analysis 16 January 2015; Test type: Superiority or Other; p = 0.0034, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.49 to 0.87]
Statistical Analysis 3: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Final Analysis 28 August 2015; Test type: Superiority or Other; p = 0.0050, Log Rank — The analysis was stratified by geographic region and metastasis classification (disease stage); Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.55 to 0.90]

3. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response was defined as a complete response or a partial response determined on two consecutive occasions ≥ 4 weeks apart. Responses were determined by Response Evaluation Criteria in Solid Tumors v1.1. A complete response was defined as the disappearance of all target lesions or the disappearance of all non-target lesions and normalization of tumor marker level. A partial response was defined as at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of the longest diameter of target lesions.
Time Frame: Baseline to the 21 July 2019 data cut-off (up to 7 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether or not study treatment was received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Number analyzed (Participants) | 247 | 248
Percentage of participants
  Primary Analysis: 9 May 2014 | 67.60 [61.39 to 73.41] | 44.80 [38.46 to 51.18]
  Post hoc Efficacy Analysis: 16 January 2015 | 69.60 [63.50 to 75.30] | 50.00 [43.60 to 56.40]
  Extended 5-Year Analysis: 21 July 2019 | 69.60 [63.49 to 75.31] | 49.60 [43.21 to 55.99]
Statistical Analysis 1: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Primary Analysis: 9 May 2014; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 22.85, 95% CI 2-sided [14.13 to 31.58]
Statistical Analysis 2: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Post hoc Efficacy Analysis: 16 January 2015; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 19.6, 95% CI 2-sided [11.0 to 28.3]
Statistical Analysis 3: Comparison: Cobimetinib + Vemurafenib vs Placebo + Vemurafenib; Extended 5-Year Analysis: 21 July 2019; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 20.00, 95% CI 2-sided [11.40 to 28.70]

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as the time from first occurrence of a documented confirmed objective response until the time of disease progression, as determined by investigator review of tumor assessments using Response Evaluation Criteria in Solid Tumors v1.1 or death from any cause during the study. Disease progression was defined as: (1) at least a 20% increase in the sum (the increase in the sum must be at least 5 mm) of diameters of target lesions, taking as reference the smallest sum during the study; (2) unequivocal progression of existing non-target lesions; or (3) the appearance of 1 or more new lesions.
Time Frame: Baseline to the 21 July 2019 data cut-off (up to 7 years, 6 months)
Population: Intent-to-treat population: All randomized participants, regardless of whether or not study treatment was received. Only participants with an objective response were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
Number analyzed (Participants) | 247 | 248
Months
  Primary Analysis: 9 May 2014 | NA [9.30 to NA] — NA = not estimable, could not be calculated due to too few events. | 7.29 [5.78 to NA] — NA = not estimable, could not be calculated due to too few events.
  Extended 5-Year Analysis: 21 July 2019: number analyzed (Participants) | 172 | 123
  Extended 5-Year Analysis: 21 July 2019 | 14.65 [12.90 to 19.30] | 9.23 [7.50 to 12.90]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of each participant's randomization into the study until their last visit until 28 days after the last dose of study drug and during extended 5-year efficacy and safety follow-up analyses (Safety data cut-off: July 2019; up to 7 years, 6 months).
Description: 1 participant was randomized in Placebo + Vem but did not receive any study treatment, 1 participant randomized in Cobi+ Vem but did not receive any study treatment, two participants were randomized in Placebo + Vem but received the Cobi+Vem.
  All-cause Mortality is reported for the ITT population, SAEs and AEs are reported for the safety population. 1 participant died after 30 days from the last dose of treatment, after crossing over from the Placebo + Vem to the Cobi+Vem arm.
Arm/Group | Cobimetinib + Vemurafenib | Placebo + Vemurafenib
All-Cause Mortality (participants affected / at risk) | 160/247 | 164/248
Serious Adverse Events (participants affected / at risk) | 105/248 | 71/245
Other Adverse Events (participants affected / at risk) | 239/248 | 236/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobimetinib + Vemurafenib (N=248) | Placebo + Vemurafenib (N=245)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 4 (8) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 1 (1) | 2 (2)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 2 (2) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 0 (0) | 4 (4)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
CHORIORETINOPATHY (Eye disorders) | 3 (5) | 0 (0)
IRIDOCYCLITIS (Eye disorders) | 0 (0) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0)
RETINAL HAEMORRHAGE (Eye disorders) | 0 (0) | 1 (1)
SEROUS RETINAL DETACHMENT (Eye disorders) | 2 (2) | 0 (0)
UVEITIS (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 3 (3) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ANTRAL VASCULAR ECTASIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OBSTRUCTION GASTRIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 2 (2)
PERIODONTAL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL POLYP (Gastrointestinal disorders) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 3 (3) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (2) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 1 (1) | 0 (0)
DEATH (General disorders) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 1 (1) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 7 (9) | 3 (3)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 2 (2)
DRUG-INDUCED LIVER INJURY (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 3 (3) | 0 (0)
SARCOIDOSIS (Immune system disorders) | 1 (2) | 0 (0)
ABDOMINAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ARTHRITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 (2) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 (2) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 1 (1) | 2 (2)
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
ERYSIPELAS (Infections and infestations) | 1 (1) | 3 (4)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 1 (1)
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1)
GASTROINTESTINAL BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GENITOURINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
GROIN ABSCESS (Infections and infestations) | 1 (2) | 0 (0)
INFECTION (Infections and infestations) | 1 (2) | 0 (0)
PNEUMONIA (Infections and infestations) | 6 (6) | 3 (3)
SEPSIS (Infections and infestations) | 1 (1) | 2 (2)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
VULVAL CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION (Infections and infestations) | 1 (1) | 0 (0)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (4) | 0 (0)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 (4) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3) | 2 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 1 (1)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 0 (0)
BLOOD CREATININE INCREASED (Investigations) | 1 (1) | 0 (0)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 1 (1)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM T WAVE ABNORMAL (Investigations) | 1 (1) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 (3) | 1 (1)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 2 (2) | 0 (0)
LIVER FUNCTION TEST INCREASED (Investigations) | 1 (1) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
ACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ADENOCARCINOMA OF COLON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
KAPOSI'S SARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 4 (4)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3)
MALIGNANT MELANOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MUCINOUS BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 2 (2) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
FACIAL PARALYSIS (Nervous system disorders) | 2 (2) | 1 (1)
FACIAL PARESIS (Nervous system disorders) | 1 (1) | 0 (0)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 2 (2) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 1 (1) | 0 (0)
MYASTHENIA GRAVIS (Nervous system disorders) | 1 (1) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 3 (3) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3) | 2 (3)
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL COLIC (Renal and urinary disorders) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1)
CERVICAL POLYP (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DERMATITIS EXFOLIATIVE GENERALISED (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DRUG REACTION WITH EOSINOPHILIA AND SYSTEMIC SYMPTOMS (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PANNICULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
RASH MORBILLIFORM (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSIVE CRISIS (Vascular disorders) | 2 (2) | 1 (1)
SUBGALEAL HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
VASCULITIS (Vascular disorders) | 1 (1) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cobimetinib + Vemurafenib (N=248) | Placebo + Vemurafenib (N=245)
ANAEMIA (Blood and lymphatic system disorders) | 51 (76) | 21 (26)
CHORIORETINOPATHY (Eye disorders) | 30 (36) | 4 (9)
VISION BLURRED (Eye disorders) | 32 (37) | 8 (9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 30 (37) | 20 (23)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 15 (17) | 18 (21)
CONSTIPATION (Gastrointestinal disorders) | 27 (37) | 29 (31)
DIARRHOEA (Gastrointestinal disorders) | 151 (311) | 84 (162)
DYSPEPSIA (Gastrointestinal disorders) | 19 (22) | 13 (15)
NAUSEA (Gastrointestinal disorders) | 108 (184) | 67 (83)
STOMATITIS (Gastrointestinal disorders) | 17 (27) | 3 (3)
VOMITING (Gastrointestinal disorders) | 69 (108) | 33 (42)
ASTHENIA (General disorders) | 51 (96) | 43 (50)
CHILLS (General disorders) | 25 (28) | 14 (17)
FATIGUE (General disorders) | 93 (137) | 83 (99)
OEDEMA PERIPHERAL (General disorders) | 38 (49) | 28 (32)
PYREXIA (General disorders) | 77 (130) | 60 (77)
CONJUNCTIVITIS (Infections and infestations) | 18 (19) | 8 (10)
FOLLICULITIS (Infections and infestations) | 19 (22) | 12 (15)
NASOPHARYNGITIS (Infections and infestations) | 23 (29) | 18 (21)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 14 (18) | 11 (15)
URINARY TRACT INFECTION (Infections and infestations) | 17 (25) | 11 (13)
SUNBURN (Injury, poisoning and procedural complications) | 37 (60) | 45 (68)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 65 (94) | 44 (48)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 64 (87) | 29 (30)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 46 (67) | 26 (30)
BLOOD BILIRUBIN INCREASED (Investigations) | 20 (29) | 17 (22)
BLOOD CHOLESTEROL INCREASED (Investigations) | 16 (19) | 10 (10)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 90 (171) | 10 (13)
BLOOD CREATININE INCREASED (Investigations) | 45 (59) | 20 (25)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 15 (30) | 8 (8)
EJECTION FRACTION DECREASED (Investigations) | 31 (46) | 12 (13)
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 12 (15) | 13 (19)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 57 (82) | 45 (61)
WEIGHT DECREASED (Investigations) | 18 (20) | 14 (17)
DECREASED APPETITE (Metabolism and nutrition disorders) | 55 (75) | 50 (55)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 13 (19) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 96 (172) | 105 (179)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 21 (30) | 15 (15)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 17 (18) | 16 (19)
MYALGIA (Musculoskeletal and connective tissue disorders) | 41 (53) | 33 (37)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 32 (51) | 40 (54)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (33) | 6 (6)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 20 (26)
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 17 (26)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 15 (15) | 21 (24)
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (26) | 30 (36)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 (25) | 33 (66)
DIZZINESS (Nervous system disorders) | 18 (18) | 7 (8)
DYSGEUSIA (Nervous system disorders) | 27 (29) | 16 (17)
HEADACHE (Nervous system disorders) | 50 (76) | 41 (50)
ANXIETY (Psychiatric disorders) | 16 (18) | 11 (12)
DEPRESSION (Psychiatric disorders) | 15 (17) | 11 (11)
INSOMNIA (Psychiatric disorders) | 19 (24) | 27 (31)
COUGH (Respiratory, thoracic and mediastinal disorders) | 28 (36) | 32 (37)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 19 (26) | 19 (23)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 22 (28)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 13 (32) | 27 (31)
ALOPECIA (Skin and subcutaneous tissue disorders) | 42 (44) | 75 (78)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 37 (47) | 22 (26)
DRY SKIN (Skin and subcutaneous tissue disorders) | 37 (40) | 42 (46)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 32 (56) | 36 (57)
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 31 (39) | 74 (130)
KERATOSIS PILARIS (Skin and subcutaneous tissue disorders) | 13 (14) | 26 (30)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 18 (23) | 9 (10)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 86 (119) | 48 (58)
PRURITUS (Skin and subcutaneous tissue disorders) | 51 (85) | 48 (54)
RASH (Skin and subcutaneous tissue disorders) | 101 (158) | 97 (121)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 37 (61) | 37 (47)
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 18 (34) | 14 (23)
HYPERTENSION (Vascular disorders) | 50 (60) | 30 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT01689519/Prot_001.pdf